CLINICAL TRIAL: NCT03620838
Title: Endometrioma Per se Versus Treatment Related Reduction in Ovarian Reserve (ERROR-2 Trial)
Acronym: ERROR2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, GÜRKAN UNCU,PROF. MD, Principal Investigator ; Prof. Dr. Gürkan Uncu, Uludag University
Other Study IDs: Uludag University
Record Dates: First submitted 2018-07-23; First posted 2018-08-08 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Ovarian Reserve; Endometrioma
MeSH Terms: conditions — Endometriosis | interventions — Contraceptives, Oral; Progesterone; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group 1: Patients with endometrioma who had at least one endometrioma >3 cm and who will not need hormonal or surgical treatment at the time of diagnosis and who will be expectantly managed
- Group 2: Patients with endometrioma who had at least one endometrioma >3 cm and who will be treated with OCP during the study period
  Interventions: Drug: oral contraceptive pill, oral progesterone
- Group 3: Patients with endometrioma who had at least one endometrioma >3 cm and who will be treated with oral progesterone during the study period
  Interventions: Drug: oral contraceptive pill, oral progesterone
- Group 4: Patients with endometrioma who had at least one endometrioma >3 cm and who will be treated with surgery short after recruitment
  Interventions: Drug: oral contraceptive pill, oral progesterone
- Group 5: The control group, who do not have endometrioma and any gynecological disorder

INTERVENTIONS:
Drug: oral contraceptive pill, oral progesterone — ovarian endometrioma cyst excision
  Other Names: surgery
  Groups: Group 2; Group 3; Group 4

SUMMARY:
The present multi-center study aimed to evaluate whether endometrioma-associated decline in ovarian reserve is progressive in the absence of an intervention and is greater in magnitude than the natural decline over time. Also the affect of endometrioma treatment modalities like surgery or medical on the ovarian reserve over time.

DETAILED DESCRIPTION:
While there is now a proven, prominent relationship between endometriosis and infertility, the exact mechanism of this relationship is still unclear. The relationship between endometriosis and infertility has been increasingly investigated in recent years. Infertility can be explained in those patients with advanced disease, which causes disturbance of the pelvic anatomy and will also prevent tubal passage, but the mechanism at the early stage of endometriosis has not yet been elucidated.

It has been shown that patients with endometriomas have low quantitative ovarian-reserve tests. It has also been shown with oocyte donation studies that endometriosis may be accompanied by a quantitative decrease in oocyte quality defects which may further adversely affect existing ovarian reserves. There are still debates as to whether the presence of endometriomas and the availability of endometriomas itself reduces the over-reserve, but there is no objective study or data on the subject.There are a number of studies that endometriosis may negatively affect the reserve, and also that surgery may cause further damage to the ovarian reserve.There is still lack of definite data for the affect of endometriomas per se and endometriomas treatment modalities ( Oral contraceptive pills (OCP) / progesterone or surgery)on the ovarian reserve over time. For this reason the investigators aimed to evaluate whether endometrioma-associated decline in ovarian reserve is progressive in the absence of any intervention and is greater in magnitude than the natural decline over time. Also the affect of endometrioma treatment modalities like surgery or medical on the ovarian reserve over time.

The study is planned as a prospective study including women with endometrioma diagnosed with ultrasonography and also healthy age matched women without endometriomas as the control group. Endometrioma patients will be divided to 4 subgroups of patients. The first group will be comprised women with endometriomas that who will not require any medical or surgical intervention, the second subgroup will be comprised from endometrioma patients will be treated with OCP during the study period, the third one will be comprised from endometrioma patients will be treated with progesterone and the last subgroup will be comprised from endometrioma patients who will be treated with surgical excision of the cyst. All of the patients with and without endometrioma will be evaluated with ultrasonography for Antral Follicle Count (AFC) and blood samples will be taken during recruitment for Anti-müllerian Hormone (AMH) values. Additional assessments will be done after 3 and 6 months after the first assessment. All the results will be statistically compared within the groups.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 40 years of age
* Who had at least one endometrioma >3 cm

Exclusion Criteria:

* İrregular periods
* Polycystic ovarian syndrome
* Pregnant patients
* Patients unable to give informed consent • Using medication which could affect ovarian function during six months before recruitment

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with endometriomas
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
AMH | 6 months
  Change from baseline Anti müllerian hormone levels at 6 months

SECONDARY OUTCOMES:
AFC | 6 months
  Change from baseline Antral follicule counts at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Uludag University Scholl of medicine, Bursa, Turkey/bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aslan K, Kasapoglu I, Kosan B, Gurbuz TB, Muzii L, Uncu G. Impact of endometrioma management strategies on ovarian reserve over the follow-up period, a prospective longitudinal study. Front Endocrinol (Lausanne). 2025 Sep 11;16:1631108. doi: 10.3389/fendo.2025.1631108. eCollection 2025. PMID 41019321